CLINICAL TRIAL: NCT06039748
Title: Diagnostic Performance of Angiography-Derived Quantitative Functional Assessment Compared to Pressure-Derived Fractional Flow Reserve and Index of Microcirculatory Resistance: The FAIR Study
Brief Title: Angiography-Derived Quantitative Functional Assessment Versus Pressure-Derived FFR and IMR: The FAIR Study
Status: Completed | Type: Observational
Sponsor: Shenzhen Raysight Intelligent Medical Technology Co., Ltd. (Industry)
Collaborators: Renmin Hospital of Wuhan University (Other); Yan'an Affiliated Hospital of Kunming Medical University (Other); Sir Run Run Shaw Hospital (Other); Jieyang People's Hospital (Other); Eighth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: The FAIR Study
Record Dates: First submitted 2023-09-10; First posted 2023-09-15 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Coronary Stenosis; Vascular Diseases; Ischemia
MeSH Terms: conditions — Coronary Artery Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Coronary Stenosis; Vascular Diseases; Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- AngioQFA
  Interventions: Other: AngioQFA

INTERVENTIONS:
Other: AngioQFA — FFR measured by pressure wire, AngioQFA computed by coronary angiographic images

SUMMARY:
Coronary angiography-derived FFR assessment (AngioQFA) is a novel technique for physiological lesion assessment based on 3-dimensional (3D) quantitative coronary angiography (QCA) and virtual hyperemic flow derived from contrast frame count without drug-induced hyperemia. The goal of this prospective, multicenter trial is to compare the diagnostic performance of AngioQFA with invasive FFR as the reference standard. The secondary purpose is to compare the diagnostic accuracies of the computational fluid dynamics (CFD)-based index of microcirculatory resistance (IMR) using wire-based IMR as the reference standard.

ELIGIBILITY:
Inclusion Criteria

* General Inclusion Criteria:

  1. Age ≥18 years.
  2. Coronary angiography is required for patients with suspected or confirmed coronary artery disease.
  3. The subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.
* Angiographic Inclusion Criteria:

  1. Diameter stenosis of 30%-90% by visual estimate
  2. Reference vessel size ≥2 mm in stenotic segment by visual estimate

Exclusion Criteria:

Patients meeting any of the following criteria will be excluded:

* General Exclusion Criteria:

  1. Subject has undergone CABG of the target vessel.
  2. Evidence of an acute myocardial infarction within one week prior to the intended procedure.
  3. Severe heart failure (NYHA≥III)
  4. Patients with other serious conditions not eligible for clinical trials, such as severe arrhythmia or tachycardia, sinus syndrome, asthma, severe chronic obstructive pulmonary disease.
  5. Serum creatinine level of >150µmol / L.
  6. Subject has known allergy to iodinated contrast agents, adenosine, or ATP.
  7. Pregnant or breastfeeding.
  8. Repeated enrollment.
  9. Any other factors that the researchers consider not suitable for diagnostic intervention or FFR and IMR detection, such as the target vessel has collateral circulation, coronary spasm, the target vessel plaque rupture resulting in myocardial infarction, or other reasons deemed unsuitable for inclusion.
* Angiographic Exclusion Criteria:

  1. Myocardial bridge or coronary artery fistula on the study lesions.
  2. The target lesion ≥50% diameter stenosis in the left main coronary artery or ostial lesions less than 3 mm to the RCA.
  3. Low-quality angiography with poor contrast agent filling or inability to detect vascular boundaries due to various reasons, vascular overlap or severe distortion of the target vessel to fully expose the lesion location is not expected to be calculated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease admitted for coronary angiography due to high risk of significant coronary stenosis
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2023-09-13 (Actual); Primary Completion 2024-01-14 (Actual); Study Completion 2024-01-14 (Actual)

PRIMARY OUTCOMES:
Diagnostic sensitivity of AngioQFA versus wire-based FFR for demonstration of coronary ischemia on a per-patient basis. | 1 hour
  Positive FFR is defined as FFR≤0.80. Positive AngioQFA is defined as AngioQFA≤0.80.
Diagnostic sensitivity of AngioIMR versus wire-based IMR for demonstration of coronary microvascular dysfunction on a per-patient basis. | 1 hour
  Positive IMR is defined as IMR≥25. Positive AngioIMR is defined as AngioIMR≥25.
Diagnostic specificity of AngioQFA versus wire-based FFR for demonstration of coronary ischemia on a per-patient basis. | 1 hour
  Negative FFR is defined as FFR>0.80. Negative AngioQFA is defined as AngioQFA>0.80.
Diagnostic specificity of AngioIMR versus wire-based IMR for demonstration of coronary microvascular dysfunction on a per-patient basis. | 1 hour
  Negative IMR is defined as IMR<25. Negative AngioIMR is defined as AngioIMR<25.

SECONDARY OUTCOMES:
Diagnostic accuracy, positive predictive value and negative predictive value of AngioQFA versus wire-based FFR for demonstration of coronary ischemia on a per-patient basis. | 1 hour
  Diagnostic accuracy, positive predictive value and negative predictive value of AngioQFA versus wire-based FFR for demonstration of coronary ischemia on a per-patient basis.
Diagnostic performance of AngioQFA in comparison to FFR on a per-vessel basis. | 1 hour
  Diagnostic performance includes sensitivity, specificity, accuracy, positive predictive value and negative predictive value.
AUC and ROC of AngioQFA Versus wire-based FFR for demonstration of ischemia on a per-vessel basis and a per-patient basis. | 1 hour
  AUC and ROC of AngioQFA Versus wire-based FFR for demonstration of ischemia on a per-vessel basis and a per-patient basis.
The consistency of AngioQFA Versus wire-based FFR for demonstration of ischemia on a per-vessel basis and a per-patient basis. | 1 hour
  The consistency of AngioQFA Versus wire-based FFR for demonstration of ischemia on a per-vessel basis and a per-patient basis.
Diagnostic accuracy, positive predictive value and negative predictive value of AngioIMR versus wire-based IMR for demonstration of coronary microvascular dysfunction on a per-patient basis. | 1 hour
  Diagnostic accuracy, positive predictive value and negative predictive value of AngioIMR versus wire-based IMR for demonstration of coronary microvascular dysfunction on a per-patient basis.
Diagnostic performance of AngioIMR in comparison to IMR on a per-vessel basis. | 1 hour
  Diagnostic performance includes sensitivity, specificity, accuracy, positive predictive value and negative predictive value.
AUC and ROC of AngioIMR Versus wire-based IMR for demonstration of coronary microvascular dysfunction on a per-vessel basis and a per-patient basis. | 1 hour
  AUC and ROC of AngioIMR Versus wire-based IMR for demonstration of coronary microvascular dysfunction on a per-vessel basis and a per-patient basis.
The consistency of AngioIMR Versus wire-based IMR for demonstration of coronary microvascular dysfunction on a per-vessel basis and a per-patient basis. | 1 hour
  The consistency of AngioIMR Versus wire-based IMR for demonstration of coronary microvascular dysfunction on a per-vessel basis and a per-patient basis.
Diagnostic sensitivity and specificity of AngioQFA and QCA DS% versus wire-based FFR for demonstration of coronary ischemia. | 1 hour
  FFR≤0.80 is defined as "positive", FFR>0.80 is defined as "negative"; DS%≥50% is defined as "positive", DS%<50% is defined as "negative".
Diagnostic accuracy of AngioQFA versus wire-based FFR for demonstration of coronary ischemia after PCI. | 1 hour
  Postoperative FFR≤0.89 was defined as "positive", FFR>0.89 is defined as "negative".
The Pearson correlation coefficient and consistency of AngioQFA Versus wire-based FFR for demonstration of ischemia on a per-vessel basis after PCI. | 1 hour
  The Pearson correlation coefficient and consistency of AngioQFA Versus wire-based FFR for demonstration of ischemia on a per-vessel basis after PCI.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Jiang, Study Director — Renmin Hospital of Wuhan University; Qiang Xue, Principal Investigator — Yan'an Affiliated Hospital of Kunming Medical University; Guosheng Fu, Principal Investigator — Sir Run Run Shaw Hospital; Jianwen Liang, Principal Investigator — The Eighth Affiliated Hospital of Sun Yat-sen University; Qiang Wu, Principal Investigator — Jieyang People's Hospital
Locations (5):
- China (5):
  - Jieyang People's Hospital, Jieyang, Guangdong
  - The Eighth Affiliated Hospital of Sun Yat-Sen University, Shenzhen, Guangdong
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Yan'an Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang